CLINICAL TRIAL: NCT05872659
Title: A Clinical Study to Evaluate the Safety and Efficacy of Human Umbilical Cord Mesenchymal Stem Cells Combined With Antiviral Therapy in the Treatment of AIDS Patients With Immune Non-responder
Brief Title: Mesenchymal Stem Cells for Immune Non-responder Patients With HIV Infection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Qilu Cell Therapy Engineering Technology Co., Ltd (Industry)
Collaborators: Shandong Public Health Clinical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSCT-A-22
Record Dates: First submitted 2023-04-11; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: AIDS Virus; Disorder of Immune Reconstitution
Keywords: HIV; mesenchymal stem cell; Immune Non-responder; CD4; AIDS; Immune reconstitution
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Participants will receive continuous antiviral therapy and saline placebo (iv, 100 mL) treatment on Day 0，Day30，Day60 and followed up for 48 weeks.
  Interventions: Other: normal saline
- Treatment group (Experimental): Participants will receive continuous antiviral therapy and Mesenchymal stem cells (1*10^6/kg subject weight, iv, 100 mL) treatment on Day 0，Day30，Day60 and followed up for 48 weeks.
  Interventions: Biological: Mesenchymal stem cells

INTERVENTIONS:
Other: normal saline — iv at D0, D30, D60
  Arms: Control group
Biological: Mesenchymal stem cells — iv at D0, D30, D60
  Arms: Treatment group

SUMMARY:
The goal of this clinical trial is to explore the effect of mesenchymal stem cell therapy on immune non-responder patients. The main questions it aims to answer are:

1. Efficacy of human umbilical cord mesenchymal stem cells combined with antiviral therapy in the treatment of AIDS patients with immune non-response.
2. Safety of human umbilical cord mesenchymal stem cells combined with antiviral therapy in AIDS patients with immune non-response.

Participants will receive CD4,CD4/CD8, and RNA viral load tests and will be randomly assigned to either saline or mesenchymal stem cell therapy.

Investigators will evaluate the safety and efficacy of mesenchymal stem cell therapy based on examination results.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) is an effective means to inhibit virus replication, increase the number of CD4+T lymphocytes and reduce mortality in HIV-infected people. However, it has been found that around 10% - 40% of patients have not achieved ideal immune function reconstruction under the condition of good viral load control and are referred to as"inadequate immunological responders" or "immune non-responders" (INRs).

A series of intervention measures have been proposed for patients with immune non-response, including growth hormone therapy, immunosuppressive therapy, cytokine therapy, traditional Chinese medicine therapy, etc., but there is no specific and effective treatment in clinical practice.

Mesenchymal stem cells (MSCs) are pluripotent stem cells with high self-renewal ability and multi-directional differentiation potential derived from mesoderm. MSCs have considerable therapeutic effects due to their migration, differentiation, immune-modulation, and regeneration abilities. The immunomodulatory effect of mesenchymal stem cells can inhibit the excessive immune activation in patients. At the same time, the paracrine effect of mesenchymal stem cells can also regulate the disordered microenvironment and promote the repair of damaged cells and tissues.

This is a randomised, placebo-controlled, clinical trial to evaluate the safety and feasibility of a 3-doses treatment regimen with MSCs (1 million cells/Kg MSCs, months 0-1-2) in HIV infected adults with immune non-response. Subjects are block randomised (1:1) to receive either MSCs (n=10), or placebo (n=10), as the control treatment. Changes in CD4+Tcount and CD4/8，adverse events, opportunistic infection signs are evaluated as determinants of safety and efficacy of MSCs. Study endpoints are measured along a follow-up period of 12 months, that includes 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection.
* ≥18 years old, gender unlimited.
* ≥12 months of continuous antiviral therapy and at least 2 viral loads (3 months or more apart) < 50 Copies/mL at screening.
* The antiviral regimen was not changed in the 12 months prior to enrollment.
* CD4+T lymphocyte count < 200 μL-1 in patients receiving antiviral therapy for more than 1 year and less than 2 years or < 350 μL-1 in patients receiving antiviral therapy for ≥ 2 years.
* Understand and sign the informed consent.

Exclusion Criteria:

* Infection with other viruses: HBV-DNA positive, HCV RNA positive, anti-Hav IgM, anti-HDV IgM and anti-HEV IgM positive and ALT >80 IU/L, anti-TP positive.
* Active and uncontrollable infection.
* Malignant tumor or tumor history.
* Complicated with abnormal function of heart, liver, lung, kidney and other major organs.
* When the laboratory test satisfies any item (WBC < 3.5*10^9/L; PLT < 80*10^9/L; HGB < 100 g/L).
* Drug dependent.
* Pregnant and lactating women.
* Severe allergic constitution, or known allergy to the study drug and its components;
* Accepting immunosuppressants or other immunomodulators (including thymosin) or systemic cytotoxic agents within 6 months prior to screening.
* Participated in other clinical studies within 3 months prior to this study.
* patients with any condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in CD4+T cell counts | Change from Baseline at 12 months
  the total CD4+T cell counts compared with CD4 T cell counts at baseline

SECONDARY OUTCOMES:
change in CD4/CD8 | Change from Baseline at 12 months
  the value of CD4/CD8 compared with CD4/CD8 value at baseline
change in RNA viral load | Change from Baseline at 12 months
  the RNA viral load compared with RNA viral load at baseline
The incidence of opportunistic infections | 12 months
  Incidence of opportunistic infections throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Chenfan liu, Principal Investigator — Shandong Public Health Clinical Center
Locations (1):
- Shandong Public Health Clinical Center, Jinan, Shandong, China